CLINICAL TRIAL: NCT02412696
Title: Placental Role in Mediating Adverse Outcomes in Obstructive Sleep Apnea
Brief Title: Positive Airway Pressure, Sleep Apnea, and the Placenta (PAP-SAP)
Acronym: PAP-SAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other); Rhode Island Hospital (Other); Women and Infants Hospital of Rhode Island (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ghada Bourjeily, MD, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1R01HD078515-01A1 (NIH)
Record Dates: First submitted 2015-01-21; First posted 2015-04-09 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea; Pregnancy; Obesity; Preeclampsia; Sleep
Keywords: placental morphology; CPAP; placental secretory function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Airway Pressure (Active Comparator): Positive airway pressure and nasal dilator strips during sleep.
  Interventions: Device: Positive Airway Pressure; Other: Nasal Dilator Strips
- Nasal Dilator Strips (Placebo Comparator): Nasal dilator strips during sleep.
  Interventions: Other: Nasal Dilator Strips

INTERVENTIONS:
Device: Positive Airway Pressure — Auto-titrating PAP + nasal dilator strips during sleep
  Arms: Positive Airway Pressure
Other: Nasal Dilator Strips — Nasal dilator strips

SUMMARY:
This study is testing the hypothesis of whether continuous positive airway pressure (CPAP) therapy improves placental histopathology and secretory function. The main aims of the study are to identify shared mechanisms between obstructive sleep apnea and preeclampsia, both common highly morbid conditions.

DETAILED DESCRIPTION:
Patients will be recruited from multiple community and hospital-based practices that care for pregnant women. Subjects will be given a physical exam, have measurements taken, answer questionnaires and then will be screened using a home sleep apnea test (HSAT) Type III device. Those diagnosed with Obstructive Sleep Apnea will then be randomized to one of two groups (below).

Both groups will have:

1. blood testing for placenta-secreted circulating markers
2. placental histopathological and immunohistochemistry examination of placental expression of markers.

Both groups will answer sleep and mood questionnaires, have blood pressure, blood glucose and activity / sleep watch monitoring and will receive an educational session on pregnancy health.

Randomization groups include:

1. Nasal dilator strips: Participants receiving nasal dilator strips will be monitored by need for refill of supplies and periodic phone calls.
2. CPAP + nasal dilator strips: Subjects randomized to positive airway pressure (PAP) therapy will receive auto-titrating PAP. Pressure requirements will be monitored remotely and pressure modified as needed. PAP adherence will be determined subjectively and objectively. This group will also receive nasal dilator strips as described above.

All subjects will receive small gift incentives such as baby-related items. Monetary incentives will also be issued at data collection points.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant snorers without obstructive sleep apnea, have a BMI >30 kg/m2 at recruitment
* >18 years of age
* <13 completed weeks of gestation (confirmed by last menstrual period or early pregnancy dating ultrasound during qualification)
* Intention to reside locally and deliver at Women and Infants Hospital of Rhode Island
* Ability to give informed consent.

Exclusion Criteria:

* Unable to meet inclusion criteria, Incompetent cervix / cerclage (likelihood of severe preterm delivery affecting study aims)
* Inability to tolerate PAP therapy
* Serious physical or mental illness or condition that would affect participation
* Drowsy driving
* Severe hypoxemia on sleep study
* Advanced cardiac disease or arrhythmias that may benefit from PAP therapy
* Chronic lung disease and / or respiratory failure.
* Twin pregnancies
* Fetuses with congenital anomalies
* Severe hypertension at enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Alterations in circulating placenta-secreted markers. | up to 6 months
  Placenta secreted markers that have been linked to preeclampsia as well as angiogenic and anti-angiogenic markers will be measured longitudinally during the course of pregnancy.
Changes in placental histopathology for markers of malperfusion and placental expression of markers | Placenta collected at time of delivery
  Placental morphology and histopathology will be examined by 3 perinatal pathologists, blinded to each other's reading and to intervention arm. Immunohistochemistry will be used to examine placental expression of certain markers.

SECONDARY OUTCOMES:
Change in 24-hour Ambulatory mean diurnal and nocturnal blood pressure measurements | Prior to randomization, then at approximately 3 months, and 6 months later
  A 24 blood pressure monitor will be used to measure changes in daytime and nighttime average blood pressure.
Change in a composite of adverse pregnancy outcomes | 8 months, delivery and 2 weeks postpartum
  Pregnancy outcomes defined as gestational hypertension, gestational diabetes and preterm birth (birth prior to 37 completed weeks of pregnancy will be analyzed as a composite outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Bourjeily, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanapo L, Bublitz MH, Bai A, Mehta N, Messerlian GM, Catalano P, Bourjeily G. Association between sleep disordered breathing in early pregnancy and glucose metabolism. Sleep. 2022 Apr 11;45(4):zsab281. doi: 10.1093/sleep/zsab281. PMID 34999843
- [Derived] Facco F. Sleep Duration, Sleep Timing, and Sleep Disordered Breathing-Associations With Obesity and Gestational Diabetes in Pregnancy. Clin Obstet Gynecol. 2021 Mar 1;64(1):196-203. doi: 10.1097/GRF.0000000000000587. PMID 33481418